CLINICAL TRIAL: NCT06993792
Title: A Master Protocol to Investigate the Efficacy and Safety of Orforglipron Tablet Once Daily Compared With Placebo in Participants With Obesity or Overweight With and Without Type 2 Diabetes
Brief Title: A Master Protocol for Orforglipron (LY3502970) in Participants With Obesity or Overweight With and Without Type 2 Diabetes
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: 27266; 2025-521098-14-00 (EU CTIS Number); J2A-MC-GZPO (Other: Eli Lilly and Company); J2A-MC-GZP1 (Other: Eli Lilly and Company); J2A-MC-GZP2 (Other: Eli Lilly and Company)
Record Dates: First submitted 2025-05-07; First posted 2025-05-29 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Obesity; Overweight; Type 2 Diabetes
MeSH Terms: conditions — Obesity; Overweight; Diabetes Mellitus, Type 2 | interventions — orforglipron

STUDY DESIGN:
Intervention Model Description: Phase 3b
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- Orforglipron Dose 1 (Study GZP1) (Experimental): Participants will receive orforglipron orally
  Interventions: Drug: Orforglipron
- Orforglipron Dose 2 (Study GZP1) (Experimental): Participants will receive orforglipron orally
  Interventions: Drug: Orforglipron
- Orforglipron Dose 3 (Study GZP1) (Experimental): Participants will receive orforglipron orally
  Interventions: Drug: Orforglipron
- Orforglipron Dose 4 (Study GZP1) (Experimental): Participants will receive orforglipron orally
  Interventions: Drug: Orforglipron
- Placebo (Study GZP1) (Placebo Comparator): Participants will receive placebo orally
  Interventions: Drug: Placebo
- Orforglipron Dose 1 (Study GZP2) (Experimental): Participants will receive orforglipron orally
  Interventions: Drug: Orforglipron
- Orforglipron Dose 2 (Study GZP2) (Experimental): Participants will receive orforglipron orally
  Interventions: Drug: Orforglipron
- Orforglipron Dose 3 (Study GZP2) (Experimental): Participants will receive orforglipron orally
  Interventions: Drug: Orforglipron
- Orforglipron Dose 4 (Study GZP2) (Experimental): Participants will receive orforglipron orally
  Interventions: Drug: Orforglipron
- Placebo (Study GZP2) (Placebo Comparator): Participants will receive placebo orally
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Orforglipron — Administered orally
  Arms: Orforglipron Dose 1 (Study GZP1); Orforglipron Dose 1 (Study GZP2); Orforglipron Dose 2 (Study GZP1); Orforglipron Dose 2 (Study GZP2); Orforglipron Dose 3 (Study GZP1); Orforglipron Dose 3 (Study GZP2); Orforglipron Dose 4 (Study GZP1); Orforglipron Dose 4 (Study GZP2)
Drug: Placebo — Administered orally
  Arms: Placebo (Study GZP1); Placebo (Study GZP2)

SUMMARY:
The purpose of this Master Protocol is to support two studies to see how well and how safely orforglipron works compared to placebo in participants who have obesity or overweight with or without type 2 diabetes. Participants will be screened for about 4 weeks, after which they will enroll into either J2A-MC-GZP1, NCT06972459 (do not have type 2 diabetes) or J2A-MC-GZP2, NCT06972472 (have type 2 diabetes).

ELIGIBILITY:
There are no specific eligibility criteria for the Master Protocol.

* See study GZP1 for eligibility criteria relevant to participants with obesity and overweight without type 2 diabetes
* See study GZP2 for eligibility criteria relevant to participants with type 2 diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2025-05-15 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Allocated to Each Study | Baseline to Week 4

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (80):
- United States (35):
  - Clinical Research Institute of Arizona (CRI) - Sun City West, Sun City West, Arizona
  - Novak Clinical Research - Tucson - North La Cholla Boulevard, Tucson, Arizona
  - Norcal Endocrinology & Internal Medicine, San Ramon, California
  - Southern California Clinical Research, Santa Ana, California
  - Care Access - Thousand Oaks, Thousand Oaks, California
  - Accel Research Sites - DeLand Clinical Research Unit, DeLand, Florida
  - Innovation Medical Research Center - Fort Lauderdale, Fort Lauderdale, Florida
  - Indago Research & Health Center, Inc, Hialeah, Florida
  - Encore Medical Research, Hollywood, Florida
  - West Orange Endocrinology P.A., Ocoee, Florida
  - Care Access - Tampa, Tampa, Florida
  - Conquest Research, Winter Park, Florida
  - Accel Research Sites - NeuroStudies Clinical Research Unit, Decatur, Georgia
  - Care Access - Decatur, Decatur, Georgia
  - Javara - Privia Medical Group Georgia - Savannah, Savannah, Georgia
  - North Georgia Clinical Research, Woodstock, Georgia
  - Solaris Clinical Research, Meridian, Idaho
  - Care Access - New Iberia, New Iberia, Louisiana
  - Endocrine and Metabolic Consultants, Rockville, Maryland
  - Javara - Privia Medical Group - Silver Spring, Silver Spring, Maryland
  - Great Lakes Research Group, Inc., Bay City, Michigan
  - Boeson Research MSO, Missoula, Montana
  - Javara - Nevada Health Centers - Carson City, Carson City, Nevada
  - The Machuca Foundation, Las Vegas, Nevada
  - University of North Carolina Medical Center, Chapel Hill, North Carolina
  - Javara - Tryon Medical Partners, Charlotte, North Carolina
  - Care Access - Fayetteville, Fayetteville, North Carolina
  - The Corvallis Clinic, P.C., Corvallis, Oregon
  - Clinical Research of Philadelphia, Philadelphia, Pennsylvania
  - Frontier Clinical Research, LLC, Smithfield, Pennsylvania
  - Velocity Clinical Research, Dallas, Dallas, Texas
  - Biopharma Informatic, LLC, Houston, Texas
  - Activian Clinical Research, Kingwood, Texas
  - Texas Valley Clinical Research (TVCR) - Mission, Mission, Texas
  - Consano Clinical Research, LLC, Shavano Park, Texas
- Argentina (6):
  - CARE - Centro de Alergia y Enfermedades Respiratorias, Buenos Aires
  - CIPREC, Buenos Aires
  - Centro Médico Viamonte, Buenos Aires
  - Instituto Centenario, CABA
  - Instituto Médico Catamarca IMEC, Rosario
  - Centro de Diagnóstico y Rehabilitación (CEDIR), Santa Fe
- China (12):
  - Xuanwu Hospital Capital Medical University, Beijing
  - Peking University Third Hospital, Beijing
  - Sichuan Provincial People's Hospital, Chengdu
  - The Second Affiliated Hospital Chongqing Medical University, Chongqing
  - Zhujiang Hospital, Guangzhou
  - The Fourth Affiliated Hospital of Harbin Medical University, Harbin
  - The Second People's Hospital of Hefei, Hefei
  - Jinan Central Hospital, Jinan
  - The First Affiliated Hospital of Henan University of Science &Technology, Luoyang Shi
  - Zhongda Hospital Southeast University, Nanjing
  - The Second Affiliated Hospital of Nanjing Medical University, Nanjing
  - The Second Hospital of Tianjin Medical University, Tianjin
- Czechia (5):
  - MUDr. Alena Vachova, České Budějovice
  - Nemocnice Cesky Krumlov, Český Krumlov
  - VASOMED Clinic, Ostrava
  - Milan Kvapil s.r.o., Diabetologicka ambulance, Prague
  - Medical Plus, Uherské Hradiště
- Germany (7):
  - InnoDiab Forschung Gmbh, Essen
  - Medizentrum Essen Borbeck, Essen
  - Diabetes Zentrum Wilhelmsburg, Hamburg
  - AmBeNet GmbH, Leipzig
  - Gemeinschaftspraxis Dr. Taeschner/Dr. Bonigut, Leipzig
  - Medicover Neuroendokrinologie, Munich
  - RED-Institut GmbH, Oldenburg
- Japan (13):
  - Hasegawa Medicine Clinic, Chitose
  - The Institute of Medical Science, Asahi Life Foundation, Chūōku
  - Tokyo-Eki Center-building Clinic, Chūōku
  - Fukuwa Clinic, Chūōku
  - Tokuyama Clinic, Mihama-ku,Chiba City
  - Medical Corporation Heishinkai ToCROM Clinic, Shinjuku-ku
  - Medical Corporation Heishinkai OCROM Clinic, Suita-shi
  - Olive Takamatsu Medical Clinic, Takamatsu
  - Shimokitazawa Tomo Clinic, Tokyo
  - Tsuchiura Medical & Health Care Center, Tsuchiura
  - Noritake Clinic, Ushiku
  - Medical Corporation Yuga Tsuruma Kaneshiro Diabetes Clinic, Yamato-shi
  - Yokohama Minoru Clinic, Yokohama
- Puerto Rico (2):
  - Puerto Rico Health and Wellness Institute, Dorado
  - Isis Clinical Research Center, Guaynabo

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/